CLINICAL TRIAL: NCT04143451
Title: Intradermal Quadrivalent Influenza Vaccine With Topical Imiquimod in Elderly & Chronic Ill Subjects, a Double-Blind Randomized Controlled Trial
Brief Title: Intradermal Influenza Vaccine With Topical Imiquimod in Elderly and Chronic Illness Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ivan FN Hung MD, Professor of Medicine, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UW 17-372
Record Dates: First submitted 2019-10-18; First posted 2019-10-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Influenza
Keywords: influenza, intradermal, imiquimod, high-dose, vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Fluzone High-Dose; Imiquimod

STUDY DESIGN:
Intervention Model Description: Double blind randomised controlled trial
Who Masked: Participant, Investigator
Masking Description: Double-blind randomization will be performed. Only the study nurse has knowledge of the type of topical treatment applied. Subjects and investigators remain blinded to the route and type of vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- IQ (Active Comparator): Year 1: a single dose ID QIV (15 µg of hemagglutinin per strain) with pre-treatment of the injected skin with imiquimod (Aldara) cream
  Year 2: randomised into 3 subgroups. Group IQ1: ID QIV (15 µg of hemagglutinin per strain) with pre-treatment of the injected skin with imiquimod (Aldara) cream Group IQ2: IM QIV (15 µg of hemagglutinin per strain with pre-treatment of the injected skin with aqueous cream. Group IQ3: ID normal saline vaccination with pre-treatment of the injected skin with imiquimod (Aldara) cream.
  Year 3: IQ1 and IQ2 same treatment as second year. IQ3 same as first year.
  Interventions: Biological: Vaxigrip tetra; Drug: Aldara 5% Topical Cream
- IM (Active Comparator): Year 1: a single dose IM QIV (15 µg of hemagglutinin per strain) with pre-treatment of the injected skin with aqueous cream
  Year 2: randomised into 3 subgroups. Group IM1: IM QIV (15 µg of hemagglutinin per strain with pre-treatment of the injected skin with aqueous cream. Group IM2: ID QIV (15 µg of hemagglutinin per strain) with pre-treatment of the injected skin with imiquimod (Aldara) cream. Group IM3: IM normal saline vaccination with aqueous cream pretreatment.
  Year 3: IM1 and IM2 same treatment as second year. IM3 same as first year.
  Interventions: Biological: Vaxigrip tetra; Drug: Aqueous cream BP
- HD (Active Comparator): Year 1: a single high-dose IM TIV (60 µg of hemagglutinin per strain) with pre-treatment of the injected skin with aqueous cream
  Year 2: Group HD1: IM QIV (60 µg of hemagglutinin per strain) with pre-treatment of the injected skin with aqueous cream. Group HD2: IM normal saline vaccination with aqueous cream pretreatment.
  Year 3: Group HD1 same treatment as second year. HD2 same as first year.
  Interventions: Biological: Fluzone high-dose; Drug: Aqueous cream BP

INTERVENTIONS:
Biological: Vaxigrip tetra — quadrivalent influenza vaccine
  Arms: IM; IQ
Biological: Fluzone high-dose — high-dose trivalent influenza vaccine
  Arms: HD
Drug: Aldara 5% Topical Cream — imiquimod cream
  Arms: IQ
Drug: Aqueous cream BP — inactive aqueous cream
  Arms: HD; IM

SUMMARY:
To compare the safety and clinical efficacy (death, overall hospitalization, hospitalization for influenza or pneumonia) of ID QIV delivered via an intradermal device with imiquimod cream pretreatment with conventional intramuscular (IM) standard dose QIV and IM high-dose TIV

DETAILED DESCRIPTION:
This is a prospective; double-blind randomized controlled study performed in the HKWC. Recruited subjects include subjects ≥50 years and adult subjects ≥18 years with chronic illness. Eligible subjects will be randomly allocated (3:3:2) into one of the three groups in the first year. Group IQ: topical 5% 250mg imiquimod ointment followed by intradermal QIV, Group IM: topical aqueous-cream followed by IM QIV and Group HD: topical aqueous-cream followed by intramuscular high-dose TIV. Hemagglutination inhibition and neutralization antibody titres will be assayed. We plan to recruit 4000 subjects, 1500 subjects in each of the IQ and IM group (500 subjects in each subgroup with 3 subgroups) and 1000 subjects for the HD group (500 subjects in each subgroup with 2 subgroups).

In the following year, the IQ and IM groups will be further randomized equally into three subgroups: IQ1, IQ2 and IQ3; IM1, IM2 and IM3; and two subgroups for HD group: HD1 and HD2. Subjects randomized to IQ1, IM1 will receive the QIV with the same topical treatment, delivery mode and vaccine as the first year and HD1 will receive the TIV with the same topical treatment, delivery mode and vaccine as the first year. Subgroup IQ2 and IM2 will be vaccinated as follow: IQ2 will receive topical aqueous-cream followed by IM QIV, IM2 will receive topical imiquimod ointment followed by ID QIV. Subgroup IQ3, IM3, HD2 will receive normal saline as the vaccine for that year, but delivered by the same mode and topical treatment. In the third year, subgroups IQ1, IQ2, IM1, IM2 and HD1 will receive the same topical treatment, delivery mode and vaccine as the second year. Subgroup IQ3, IM3 and HD2 will receive the same topical treatment, delivery mode and vaccine as the first year.

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include subjects ≥50 years or adult subjects ≥18 years with chronic illness attending GOPD or SOPD in HKWC.
2. All subjects/ next of kin give written informed consent.
3. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Have a recent history (documented, confirmed or suspected) of a flu-like disease within a week of vaccination.
3. Have a known allergy to eggs or other components of the study vaccines (including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein), or history of any anaphylaxis, serious vaccine reactions, to any excipients.
4. Have an active neoplastic disease or a history of active hematologic malignancy.

4. Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.

6. Have known active human immunodeficiency virus (HIV) infection. 7. Received an agent on clinical trial (vaccine, drug, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study. Unwilling to refuse participation in another clinical study through the end of this study.

8. Tympanic temperature ≥ 38°C within 3 days of intended study vaccination 9. Have a history of alcohol or drug abuse in the last 5 years. 10. Have a history of Guillain-Barré Syndrome. 11. Pregnant during the study period. 12. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 years
  death rate
Overall hospitalisation | 3 years
  hospitalisation rate for all diagnosis
Hospitalisation for influenza | 3 years
  hospitalisation rate with microbiological confirmation of influenza
Hospitalisation for pneumonia | 3 years
  hospitalisation rate with a clinical diagnosis of pneumonia

SECONDARY OUTCOMES:
immediate adverse events | 5 minutes post vaccination
  immediate adverse events
adverse events | 7 days post vaccination
  Local: redness, swelling, induration, pain and ecchymosis. Redness, swelling, and induration will be graded based on size: Grade 1, under 20mm; Grade 2, 20-50mm. Pain will be graded as follows: Grade 1, pain on touch, Grade 2, pain when arm is moved Systemic: fever, headache, malaise, myalgia, arthralgia and severe adverse events.
immunogenicity | at 21 days, 6 months and 1 year after each vaccination
  GMT, seroconversion rate, seroprotection rate and GMT fold increase by HI and MN assays on day, 21, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No